CLINICAL TRIAL: NCT04302389
Title: Single Arm Trial of a Multi-component Commercial Digital Weight Loss Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Principal Investigator, Sherry Pagoto, Professor, University of Connecticut
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H20-0030
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: This project includes a one-arm trial to evaluate WW's new lifestyle modification program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle Modification Program (Experimental): This 6-month intervention includes the use of three components: WW's mobile app, virtual workshops, and a private online community. The WW Program involves: self-monitoring of weight, dietary intake, and physical activity; making dietary changes; increasing physical activity; shifting to a more helpful mindset; and learning behavioral strategies to manage these goals. Each week, participants will set goals and weigh-in with a coach via virtual workshop. Participants will be encouraged to use the app and private online community daily and attend weekly virtual workshops. The weekly virtual workshop led by a trained WW Coach features a behavior change technique and enables the participant to practice it to support their goals. These are actionable techniques and strategies that are grounded in scientific research.
  Interventions: Behavioral: myWW App, Virtual Workshops, and Private Facebook Group

INTERVENTIONS:
Behavioral: myWW App, Virtual Workshops, and Private Facebook Group — The 6-month intervention includes the use of WW's mobile app, weekly virtual workshops, and a private online community. Participants are given a personalized food plan based on expert healthy eating guidelines and the latest nutritional science, an activity plan designed to promote regular physical activity and techniques to help shift members towards a helpful mindset for lasting change all within the WW app. Participants will attend weekly virtual workshops led by an expert WW Coach. The coach will help with goal setting, overcoming setbacks, and follow-up on progress toward goals each week. Participants will be encouraged to participate in a private Facebook group that gives participants an opportunity to receive motivational support from each other. Participants can post about their journey through photos, videos, and comments.

SUMMARY:
The goal of the proposed research project is to evaluate the acceptability and efficacy of an online multicomponent commercial weight loss program and to understand the relationship between program engagement and weight loss and health outcomes.

DETAILED DESCRIPTION:
Technology is changing the opportunities to deliver behavioral weight loss programs and providing a way to extend their reach to wider audiences. Commercial programs that were once completely delivered via in person meetings at brick-and-mortar businesses are now expanding to virtual programs. WW (formerly known as Weight Watchers) is an industry leader and one of few commercial programs that has significant evidence for efficacy on weight loss. Their program currently includes a mobile app - that helps people follow the WW Program, rewards for consistent tracking and achieving milestones, an online community to connect with other users, and a 24/7 text chat with coaches.

Previous research by the investigators and others reveals that greater engagement in an online group-based weight loss program is associated with greater weight loss. We have found that an online group coaching program paired with a calorie tracking mobile app is effective at producing weight loss. WW is testing a new comprehensive program that involves an updated program paired with virtual workshops that offer actionable behavior change techniques for members, led by a trained WW coach. They have agreed to fund us to perform a one-arm trial of their new comprehensive program that includes a holistic approach to healthy lifestyle (activity, diet, and mindset). Findings will inform the continued development of this program. Our aims are as follows: 1) To examine the preliminary outcomes and acceptability of a multicomponent online commercial weight loss program that includes a mobile app, incentives for tracking, weekly virtual workshops, and an online community. Preliminary outcome is defined as weight change from baseline to 3 and 6-months. Secondary preliminary outcomes include changes in diet quality, physical activity, quality of life, sleep quality, and food cravings from baseline to 6 months. Acceptability of each program component and the overall program will be evaluated at 6 months. 2) To examine whether greater app use, greater engagement in the online community, and engagement with a higher number of peers (in the online community) predict greater weight loss at 3- and 6-months. 3) To examine the associations between total use of program components (and each individual program component) and change in weight. We hypothesize that greater use of program components (individually and total) will predict greater weight loss.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old.
2. BMI 25-45 kg/m2.
3. Has Wi-Fi connectivity at home
4. Able to participate in the study in English.
5. Self-reported desire to lose weight.
6. Willing to follow recommendations required by study protocol.
7. Willing to include demographic information (e.g., ethnicity, income and education)
8. Lives in the United States

Exclusion Criteria:

1. Pregnant, lactating, or plans to become pregnant during study period.
2. Bipolar disorder, substance abuse, psychosis, bulimia, binge eating disorder, or severe depression.
3. Had bariatric surgery or plans to have any surgery during the study
4. Unable to make dietary changes or increase physical activity.
5. Unable to walk ¼ mile unaided without stopping
6. Smoker or use nicotine vape daily.
7. Participants that are currently, or within the last 6 months, trying to lose weight via a structured weight-loss program (e.g., at a medical center, university, commercial programs)
8. Participants who were a member of WW within the past 12 months.
9. Participants who are involved in any other research studies at this time.
10. Weight loss of ≥ 5 kg in the previous 6 months.
11. Reported health problems that make weight loss or unsupervised exercise unsafe or unreasonable (e.g., chronic pain, orthopedic limitations, heart problems).
12. Untreated thyroid disease or any changes (type or dose) in thyroid medication in last 6 months.
13. Taking any prescription medication with known effects on appetite or weight (e.g., oral steroids, weight loss medications such as Qysmia, Contrave, etc.) with the exception of subjects on a stable dose of SSRIs for 6 months.
14. Chronic/inflammatory gastrointestinal disorders (irritable bowel syndrome is acceptable).
15. History of heart problems (e.g., angina, bypass surgery, myocardial infarction, etc.) within previous 6 months.
16. Diagnosis of type 1 or type 2 diabetes.
17. Major surgery within the previous 6 months.
18. Presence of implanted cardiac defibrillator or pacemaker.
19. History of cancer within past 5 years or current treatment for cancer (completely resected basal or squamous cell carcinoma acceptable if treatment completed more than 6 months prior to enrollment).
20. Meets criteria for severe depression on the PHQ-9 (score of >20) or endorsement of "Thoughts that you would be better off dead, or of hurting yourself in some way".
21. Hospitalization for psychiatric disorders during the past 12 months.
22. Not willing to sign an NDA; or indicated they do not want to agree to NDA's terms.
23. Unable to attend any virtual workshop meeting times.
24. Does not have an iPhone.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Pagoto, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu R, Bannor R, Cardel MI, Foster GD, Pagoto S. How much food tracking during a digital weight-management program is enough to produce clinically significant weight loss? Obesity (Silver Spring). 2023 Jul;31(7):1779-1786. doi: 10.1002/oby.23795. Epub 2023 Jun 4. PMID 37271576

RESULTS

PARTICIPANT FLOW:
Groups:
- Lifestyle Modification Program: This 6-month intervention includes the use of three components: WW's mobile app, virtual workshops, and a private online community. The WW Program involves: self-monitoring of weight, dietary intake, and physical activity; making dietary changes; increasing physical activity; shifting to a more helpful mindset; and learning behavioral strategies to manage these goals. Each week, participants will set goals and weigh-in with a coach via virtual workshop. Participants will be encouraged to use the app and private online community daily and attend weekly virtual workshops. The weekly virtual workshop led by a trained WW Coach features a behavior change technique and enables the participant to practice it to support their goals. These are actionable techniques and strategies that are grounded in scientific research.
  myWW App, Virtual Workshops, and Private Facebook Group: The 6-month intervention includes the use of WW's mobile app, weekly virtual workshops, and a private online community. Participants are given a personalized food plan based on expert healthy eating guidelines and the latest nutritional science, an activity plan designed to promote regular physical activity and techniques to help shift members towards a helpful mindset for lasting change all within the WW app. Participants will attend weekly virtual workshops led by an expert WW Coach.
Period: Overall Study
Arm/Group | Lifestyle Modification Program
Started | 153
Completed | 141
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107
  Male | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 134
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 107
  More than one race | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 153
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.77 (5.02)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Days Diet Tracking Feature Was Used in App
Description: Percent of days participants used the diet tracking feature in the WW app during the intervention to track their daily food intake. A day of use will be defined as a day where participants tracked any food item in the WW app.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent of days of tracking food
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 153
percent of days of tracking food | 39.1 (30.8)

2. Primary Outcome: Intervention Acceptability
Description: Percent of participants who agree or strongly agree that the program made them feel healthier.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 140
Participants | 102

3. Primary Outcome: Percent Change in Weight From Baseline to 3 Months
Description: Weight was measured using a smart scale at baseline and at the three month assessment.
Time Frame: Baseline to 3-months
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 153
Percent change | -8.19 (7.51)
Statistical Analysis 1: Comparison: Lifestyle Modification Program; This was a within-subject comparison at two timepoints (baseline, 3 months); Test type: Other; p < 0.001, t-test, 2 sided

4. Primary Outcome: Weight Change in Pounds From Baseline to 6 Months
Description: Weight will be measured using a smart scale at all assessments. Weight change will be calculated as weight at 6 months in pounds minus baseline weight in pounds. Lower values mean more weight loss.
Time Frame: Baseline to 6-months
Measure: Mean (Standard Deviation); unit: weight change in pounds
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 153
weight change in pounds | -9.72 (10.78)

5. Primary Outcome: Number of Days Physical Activity Tracking Feature Was Used in App
Description: Number of days participants used the physical activity feature in the WW app during the intervention. A day of use will be defined as any day in which any physical activity was logged. Total days possible = 168 days.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 153
days | 106.37 (73.22)

6. Primary Outcome: Number of Weekly Virtual Workshops Attended
Description: Number of weekly workshops attended by participants during the program. During the 6-month intervention, there were a total of 24 weekly workshops.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: number of weekly workshops attended
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 153
number of weekly workshops attended | 9.68 (7.16)

7. Primary Outcome: Number of Weekly Check Ins Attended
Description: Number of weekly check ins completed by participants during the program. During the 6-month intervention, there were 24 opportunities for weekly check ins. Higher numbers mean more weekly check ins were completed.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: number of weekly check-ins attended
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 153
number of weekly check-ins attended | 11.91 (7.63)

8. Primary Outcome: Number of Weeks Participants Engaged in the Private, Online Community
Description: All posts, comments, and reactions made in the Facebook group were captured using Grytics for Facebook each of the 24 weeks of the intervention. Participants were considered engaged with the intervention by making at least one post, one comment, and/or one reaction (e.g., like) during the intervention week. Values could range from 0 to 24 weeks with higher numbers indicating more frequent engagement in the intervention.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: number of weeks a participant engaged
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 153
number of weeks a participant engaged | 6.03 (7.03)

9. Primary Outcome: Weight Change in Pounds From Baseline to 3 Months
Description: Weight will be assessed via digital scales provided to participants. Weight change will be calculated by subtracting weight in pounds at 3 months from baseline weight. Lower values indicate greater weight loss in pounds.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: weight in pounds
Groups:
- Lifestyle Modification Program: This 6-month intervention includes the use of three components: WW's mobile app, virtual workshops, and a private online community. The WW Program involves: self-monitoring of weight, dietary intake, and physical activity; making dietary changes; increasing physical activity; shifting to a more helpful mindset; and learning behavioral strategies to manage these goals. Each week, participants will set goals and weigh-in with a coach via virtual workshop. The weekly virtual workshop led by a trained WW Coach.
  myWW App, Virtual Workshops, and Private Facebook Group: The 6-month intervention includes the use of WW's mobile app, weekly virtual workshops, and a private online community. Participants are given a personalized food plan based on expert healthy eating guidelines and the latest nutritional science, an activity plan designed to promote regular physical activity and techniques to help shift members towards a helpful mindset for lasting change all within the WW app. Participants will attend weekly virtual workshops led by an expert WW Coach. The coach will help with goal setting, overcoming setbacks, and follow-up on progress toward goals each week. Participants will be encouraged to participate in a private Facebook group that gives participants an opportunity to receive motivational support from each other. Participants can post about their journey through photos, videos, and comments.
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 153
weight in pounds | -8.19 (7.51)

10. Primary Outcome: Percent Weight Change From Baseline to 6 Months
Description: Weight is assessed via digital scales provided to participants. Percent weight change will be calculated by subtracting 6 month weight in pounds from baseline weight in pounds, dividing by baseline weight in pounds, and then multiplying this number by 100. Lower values indicated greater weight loss.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent weight change
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 153
percent weight change | -5.05 (5.59)

11. Secondary Outcome: Change in Fruit Intake Score
Description: At baseline and 6 months, participants completed the National Health Interview Survey Five-Factor Screener, which contains 19 items that assess the consumption frequency (measured on a scale ranging from 0=never to 5=≥5 times per day) of different food groups, including fruit intake. 1 assessed fruit intake. Change in fruit intake score was calculated by subtracting 6 month values from baseline values. Higher change scores indicate greater increases in fruit intake.
Time Frame: Baseline to 6-months
Measure: Mean (Standard Deviation); unit: scores on scale of 0-5
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 132
scores on scale of 0-5 | .18 (.82)

12. Secondary Outcome: Change in Physical Activity
Description: Changes in physical activity will be measured from baseline to 6-months using the Global Physical Activity Questionnaire (GPAQ). The GPAQ has questions assessing activity at work, travel to and from places, and recreational activities. The number of minutes spent on each activity is assigned a METs value to determine level of energy expenditure. The higher the METs value the higher the activity level.
Time Frame: Baseline to 6-months
Measure: Mean (Standard Deviation); unit: METs
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 141
METs | 783.95 (3611.88)

13. Secondary Outcome: Changes in Quality of Life
Description: Changes in weight related quality of life will be measured from baseline to 6-months using the Impact of Weight on Quality of Life-Lite. This is a 31-item measure assessing physical function (11 items), self-esteem (7 items), sexual life (4 items), public distress (5 items), and work (4 items). Scores range from 0-100, with 100 representing the best quality of life. Change was calculated by subtracting 6 month scores from baseline scores. Higher values indicate greater increases in quality of life.
Time Frame: Baseline to 6-months
Measure: Mean (Standard Deviation); unit: score on scale of 0-100
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 141
score on scale of 0-100 | 6.63 (11.51)

14. Secondary Outcome: Changes in Sleep Quality
Description: Changes in sleep quality will be measured from baseline to 6-months using the Pittsburgh Sleep Quality Index. This measure contains 10 items to assess sleep quality with a score possible score of 0 - 21. Lower scores represent better the sleep quality (< 5 is associated with good sleep quality; > 5 is associated with poor sleep quality. Change in sleep quality was calculated by subtracting 6 month scores from baseline scores. Lower values indicate improvements in sleep quality.
Time Frame: Baseline to 6-months
Measure: Mean (Standard Deviation); unit: score on a 0-21 scale
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 141
score on a 0-21 scale | -.56 (2.56)

15. Secondary Outcome: Changes in Food Cravings
Description: Changes in food cravings will be measured from baseline to 6-months using the Food Craving Inventory. This inventory includes 28 foods that are scored based on level of craving ranging in answers from 1 (Never) to 5 (Always) for each. A mean is calculated across the 28 items. Scores then would range from a minimum of 1 to a maximum of 5. Higher scores indicate more frequent cravings. Change was calculated by subtracting 6 month scores from baseline scores. Higher scores indicate greater increases in food cravings.
Time Frame: Baseline to 6-months
Measure: Mean (Standard Deviation); unit: mean scores on a scale
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 141
mean scores on a scale | -.42 (.52)

16. Secondary Outcome: Changes in Hunger
Description: Changes in hunger will be measured from baseline to 6-months using the Hunger VAS (Visual Analogue Scale). This one-question measure asks "How hungry did you feel over the past week" and is composed of a slider with words anchored at each end describing the extremes (Not at all hungry, Extremely hungry). Participants rated their hunger over the past week using a slider on a visual analog scale ranging from 0=not at all hungry to 100=extremely hungry. Change in hunger was then calculated by subtracting the hunger score at 6 months from the hunger score at baseline. Higher values indicate increases in hunger over time and lower values indicate decreases in hunger over time.
Time Frame: Baseline to 6-months
Measure: Mean (Standard Deviation); unit: score on a 0-100 scale
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 141
score on a 0-100 scale | -13.02 (22.23)

17. Secondary Outcome: Changes in Positive Behavioral Automaticity
Description: Changes in behavioral automaticity will be measured using the Self-Report Behavioral Automaticity Index (SRBAI). This 4-item measure assesses whether Behavior X is something... "I do automatically", "I do without having to consciously remember", "I do without thinking", and "I start doing before I realize I'm doing it". Items are scored using a 7-point Likert scale ranging from strongly disagree to strongly agree. A mean score was calculated for each behavior. Then, mean scores were calculated for the 7 healthy behaviors to produce a positive behavioral automaticity score which could range from 1 to 7. Change in positive behavioral automaticity was then calculated by subtracting the 6 month value from the baseline value. Higher scores indicate greater behavioral automaticity for healthy behaviors.
Time Frame: Baseline to 6-months
Measure: Mean (Standard Deviation); unit: score on a scale of 1-7
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 141
score on a scale of 1-7 | .86 (1.09)

18. Secondary Outcome: Changes in Self-Compassion
Description: Changes in self-compassion will be measured using the Self-Compassion Scale. This is a 26-item measure of self-compassion that consists of six subscales: self-kindness, self-judgement, common humanity, isolation, mindfulness, and over-identified. Items were rated a scale ranging from 1=almost never to 5=almost always. Subscales are computed by calculating the mean of subscale item responses. A total self-compassion score can be obtained by reverse scoring the negative subscale items (self-judgement, isolation, and over-identification) and computing a grand mean of all six subscale means. The total possible scores range from 1-5. Then to calculate change in self-compassion, we subtracted the 6 month value from the baseline value. Higher scores mean greater increases in self-compassion over time.
Time Frame: Baseline to 6-months
Measure: Mean (Standard Deviation); unit: score on a scale from 1-5
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 141
score on a scale from 1-5 | .09 (.56)

19. Secondary Outcome: Change in Well-being
Description: Changes in well-being will be measured using the WHO-5 Well Being Index (0-100 score where higher scores mean greater well-being). Change in well-being was then calculated by subtracting the 6 month score from the baseline score. Higher values indicate increases in well-being over time.
Time Frame: Baseline to 6-months
Measure: Mean (Standard Deviation); unit: score on a 0-100 scale
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 141
score on a 0-100 scale | 5.96 (15.36)

20. Secondary Outcome: Change in Vegetable Intake Score
Description: At baseline and 6 months, participants completed the National Health Interview Survey Five-Factor Screener, which contains 19 items that assess the consumption frequency (measured on a scale ranging from 0=never to 5=≥5 times per day) of different food groups, including fruits and vegetables. 1 assessed vegetable intake. Change in vegetable intake score was calculated by subtracting 6 month values from baseline values. Higher change scores indicate greater increases in vegetable intake.
Time Frame: baseline to 6 months
Measure: Mean (Standard Deviation); unit: scores on scale of 0-5
Groups:
- Lifestyle Modification Program: This 6-month intervention includes the use of three components: WW's mobile app, virtual workshops, and a private online community. The WW Program involves: self-monitoring of weight, dietary intake, and physical activity; making dietary changes; increasing physical activity; shifting to a more helpful mindset; and learning behavioral strategies to manage these goals. Each week, participants will set goals and weigh-in with a coach via virtual workshop. The weekly virtual workshop is led by a trained WW Coach.
  myWW App, Virtual Workshops, and Private Facebook Group: The 6-month intervention includes the use of WW's mobile app, weekly virtual workshops, and a private online community. Participants are given a personalized food plan based on expert healthy eating guidelines and the latest nutritional science, an activity plan designed to promote regular physical activity and techniques to help shift members towards a helpful mindset for lasting change all within the WW app. Participants will attend weekly virtual workshops led by an expert WW Coach. The coach will help with goal setting, overcoming setbacks, and follow-up on progress toward goals each week. Participants will be encouraged to participate in a private Facebook group that gives participants an opportunity to receive motivational support from each other. Participants can post about their journey through photos, videos, and comments.
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 132
scores on scale of 0-5 | .16 (.7)

21. Secondary Outcome: Change in Salad Intake Score
Description: At baseline and 6 months, participants completed the National Health Interview Survey Five-Factor Screener, which contains 19 items that assess the consumption frequency (measured on a scale ranging from 0=never to 5=≥5 times per day) of different food groups, including fruits and vegetables. 1 assessed salad intake. Change in salad intake score was calculated by subtracting 6 month values from baseline values. Higher change scores indicate greater increases in salad intake.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: scores on scale of 0-5
Groups:
- Lifestyle Modification Program: This 6-month intervention includes the use of three components: WW's mobile app, virtual workshops, and a private online community. The WW Program involves: self-monitoring of weight, dietary intake, and physical activity; making dietary changes; increasing physical activity; shifting to a more helpful mindset; and learning behavioral strategies to manage these goals. Each week, participants will set goals and weigh-in with a coach via virtual workshop. The weekly virtual workshop will be led by a trained WW Coach.
  myWW App, Virtual Workshops, and Private Facebook Group: The 6-month intervention includes the use of WW's mobile app, weekly virtual workshops, and a private online community. Participants are given a personalized food plan based on expert healthy eating guidelines and the latest nutritional science, an activity plan designed to promote regular physical activity and techniques to help shift members towards a helpful mindset for lasting change all within the WW app. Participants will attend weekly virtual workshops led by an expert WW Coach. The coach will help with goal setting, overcoming setbacks, and follow-up on progress toward goals each week. Participants will be encouraged to participate in a private Facebook group that gives participants an opportunity to receive motivational support from each other. Participants can post about their journey through photos, videos, and comments.
Arm/Group | Lifestyle Modification Program
Number analyzed (Participants) | 132
scores on scale of 0-5 | .18 (.53)

ADVERSE EVENTS:
Time Frame: 6 months
Description: The definition does not differ.
Arm/Group | Lifestyle Modification Program
All-Cause Mortality (participants affected / at risk) | 0/153
Serious Adverse Events (participants affected / at risk) | 13/153
Other Adverse Events (participants affected / at risk) | 0/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle Modification Program (N=153)
heart attack (Cardiac disorders) | 1 (1) — Participant reported via email on 3/30 that she was admitted to the hospital due to having a heart attack. We received the email morning of 3/31. This happened prior to the start date of the study. Stents were placed in 2 vessels.
broken leg (Musculoskeletal and connective tissue disorders) | 1 (1) — Participant broke leg in a motorcycle accident and was admitted to the hospital and had surgery to insert a pin to support the bone. Participant was casted and referred to physical therapy.
multiple sclerosis flare up (Musculoskeletal and connective tissue disorders) | 1 (1) — Participant reported nerve pain in the face (trigeminal neuralgia) and went to a neurologist for care. Treatment involved medication.
diverticulitis (Gastrointestinal disorders) | 1 (1) — Participant reported a diagnosis of diverticulitis on the AE form. Participant went to doctor and was put on antibiotics.
Hernia (Musculoskeletal and connective tissue disorders) | 1 (1) — Participant indicated on the AE form that they had hernia surgery.
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) — Participant indicated that they fell off of a cliff while hiking on vacation. They were taken to the hospital and had soft tissue injuries and lacerations treated.
hysterectomy (Reproductive system and breast disorders) | 1 (1) — Participant stated on AE form that they had an emergency outpatient hysterectomy. They were on bedrest for 2 weeks during recovery.
sarcoidosis (Blood and lymphatic system disorders) | 1 (1) — Participant indicated on AE form that they discovered swollen lymph nodes and were diagnosed with sarcoidosis. They received a lymph node biopsy and were put on hydroxychloroquine.
Sarcoidosis flare up (Blood and lymphatic system disorders) | 1 (1) — Participant indicated on the 6 month survey they had a sarcoidosis flare up that affected their energy level. They were under their physician's care.
tardive dyskinesia (Musculoskeletal and connective tissue disorders) | 1 (1) — Participant indicated on the 3 month survey that due to the medication they were taking they were diagnosed with tardive dyskinesia.
thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Participant said they noticed their neck was slightly enlarged. They went to their doctor and was given a biopsy and a lobectomy which revealed stage 1 papillary thyroid cancer. The rest of the thyroid was removed. They are now cancer free.
eosinophilic gastrointestinal disease (EGID) (Gastrointestinal disorders) | 1 (1) — Participant withdrew from the study after being diagnosed with EGID. Their doctor referred them to dietary counseling.
tubal ligation (Reproductive system and breast disorders) | 1 (1) — Participant had an IUD embedded and had to have it surgically removed along with receiving a tubal ligation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT04302389/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT04302389/SAP_001.pdf
  • Informed Consent Form (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT04302389/ICF_002.pdf